CLINICAL TRIAL: NCT03161873
Title: Cycle and Pregnancy Monitoring With Wearable Sensor Technology (AVA)
Acronym: SUSAVA
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Ava AG (Industry); CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Other Study IDs: S_US_Ava
Record Dates: First submitted 2017-05-09; First posted 2017-05-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Fertility Disorders; Early Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- avaOnly: Participants will measure with Ava bracelet and determine ovulation with a home (luteinizing hormone) LH urine test
  Interventions: Device: Ava
- avaSaliva: Participants will measure with Ava bracelet and determine ovulation with a home LH urine test. In addition participants will collect saliva for the measurements of estrogen and progesterone.
  Interventions: Device: Ava
- avaSalivaUS: Participants will measure with Ava bracelet and determine ovulation with a home LH urine test. In addition participants will collect saliva for the measurements of estrogen and progesterone. Moreover ultrasound will be used to observe the day at which the ovum is released.
  Interventions: Device: Ava
- avaBBT: Participants will measure with Ava bracelet and determine ovulation with a home LH urine test. In addition, participants will measure their basal body temperature (BBT) daily.
  Interventions: Device: Ava

INTERVENTIONS:
Device: Ava — Ava is a fertility monitoring bracelet that collects various physiological parameters

SUMMARY:
In this study physiological data is measured using wearable sensors as well as hormonal and ultrasound measurements of growing follicles/ ovulation in a group of endocrinologically healthy women with regular cycles, who aim for a spontaneous pregnancy. These women were recruited to generate reliable data on changes of the measured physiological parameters in a healthy menstrual cycle, as well as to evaluate physiological changes associated with early pregnancy.

All pregnancies beginning during the study period are to be monitored to their natural end, in order to evaluate how the same nine physiological parameters are changing during pregnancy, how strong the variations of the parameters during pregnancy are, and whether they could be associated with early onsets of pregnancy complications such as premature birth or pre-eclampsia. This will be highly valuable to develop study protocols for the specific evaluation of the screening potential of pregnancy complications.

ELIGIBILITY:
Inclusion Criteria:

* women aged 20-40 years
* regular menstrual cycle (28 days+/-)
* no hormonal therapy
* German-speaking
* written informed consent to participate in the study

Exclusion Criteria:

* any health-related issues that may affect menstrual cycle
* any consumption of medication or other substances that may affect the menstrual cycle or any of the physiological parameters investigated
* frequent travel between time zones
* sleeping disorders
* unsuccessfully trying to conceive for > 12 months

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study we want to conduct measurements of physiological data as well as hormonal and ultrasound measurements of growing follicles/ ovulation in a group of endocrinologically healthy women with a regular cycle, who aim for a spontaneous pregnancy. We choose these women to generate reliable data on changes of the measured physiological parameters in a healthy menstrual cycle, as well as to evaluate physiological changes associated with the initiation of pregnancy.
  We want to continue measurements in all pregnancies beginning during the study period to evaluate how the same nine physiological parameters are changing during pregnancy, how strong the variations of the parameters during pregnancy are, and whether they could be associated with early onsets of pregnancy complications such as premature birth or preeclampsia. This will be highly valuable to develop study protocols for the specific evaluation of the screening potential of one of the pregnancy complications.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Correlation between the physiology and the menstrual cycle dynamics | November 2016 - November 2020
  Correlation between a the following physiological parameters (individually or in combination), pulse rate, respiration, skin conductance response, sleep duration and quality, and skin perfusion with the menstrual cycle dynamics

SECONDARY OUTCOMES:
Correlation between the physiology measured using a wearable device and the occurrence of pregnancy | November 2016 - November 2020
  Correlation between the following physiological parameters (individually or in combination), pulse rate, respiration, skin conductance response, sleep duration and quality, and skin perfusion with the occurrence of pregnancy.
Correlation between physiology and pregnancy complications | November 2016 - November 2020

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Leeners, Prof, Principal Investigator — University of Zurich
Locations (1):
- Clinic for Reproductive Endocrinology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No